CLINICAL TRIAL: NCT05338489
Title: A 2-Part, Open-Label, Fixed-Sequence Study to Evaluate the Effects of Multiple Doses of Itraconazole and Rifampin on the Single-Dose Pharmacokinetics of LOXO-292 in Healthy Adult Subjects
Brief Title: A Study of Effects of Itraconazole and Rifampin on Selpercatinib (LY3527723) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17751; J2G-OX-JZJP (Other: Eli Lilly and Company); LOXO-RET-18014 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-04-19; First posted 2022-04-21 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — selpercatinib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole (Experimental): Participants received a single oral dose of 160 milligrams (mg) selpercatinib on Day 1 of Period 1.
  In Period 2, participants received an oral dose of 200 mg itraconazole administered once daily (QD) for 11 consecutive days (Days -4 to 7) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 of Period 2.
  There was a washout period of at least 7 days between the dose of selpercatinib in Period 1 and the first dose of itraconazole in Period 2.
  Interventions: Drug: Selpercatinib; Drug: Itraconazole
- Part 2 - 160 mg Selpercatinib + 600 mg Rifampin (Experimental): Participants received a single oral dose of 160 mg selpercatinib on Day 1 of Period 1.
  In Period 2, participants received an oral dose of 600 mg rifampin administered QD for 16 consecutive days (Days 1 to 16) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 and Day 10 of Period 2.
  There was a washout period of at least 7 days between the dose of selpercatinib in Period 1 and the first dose of rifampin and selpercatinib in Period 2.
  Interventions: Drug: Selpercatinib; Drug: Rifampin

INTERVENTIONS:
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292
Drug: Itraconazole — Administered orally.
  Arms: Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole
Drug: Rifampin — Administered orally.
  Arms: Part 2 - 160 mg Selpercatinib + 600 mg Rifampin

SUMMARY:
The main purpose of this study is to assess the effect of itraconazole and rifampin on how fast selpercatinib gets into the blood stream and how long it takes the body to remove it when administered in healthy participants. Information about safety and tolerability will be collected. The study is conducted in two parts and it will last up to 54 days (part 1) and 59 days (part 2), respectively, inclusive of screening period.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential who are agreeable to take birth control measures until study completion
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Have previously participated or withdrawn from this study
* Have or used to have health problems or laboratory test results or ECG readings that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Had blood loss of more than 500 milliliters (mL) within the previous 30 days of study screening
* Require treatment with inducers or inhibitors of cytochrome P450 (CYP) CYP3A within 14 days before the first dose of study drug through the end of Period 2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2018-07-28 (Actual); Study Completion 2018-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 - 160 mg Selpercatinib + 600 mg Rifampin
Started | 12 | 12
Received at Least One Dose of Study Drug | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 - 160 mg Selpercatinib + 600 mg Rifampin
Started | 12 | 12
Received at Least One Dose of Study Drug | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole: Participants received a single oral dose of 160 mg selpercatinib on Day 1 of Period 1.
  In Period 2, participants received an oral dose of 200 mg itraconazole administered QD for 11 consecutive days (Days -4 to 7) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 of Period 2.
  There was a washout period of at least 7 days between the dose of selpercatinib in Period 1 and the first dose of itraconazole in Period 2.
- Total: Total of all reporting groups
Arm/Group | Part 1 - 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 - 160 mg Selpercatinib + 600 mg Rifampin | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (7.81) | 37.8 (7.15) | 39.1 (7.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 10 | 9 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Description: PK: AUC0-t of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: (contd.) Part 2, Period 2: (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post dose; (Day 10) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram *hour per milliliter (ng*h/mL)
Groups:
- Part 1 Period 1: 160 mg Selpercatinib; Part 2 Period 1: 160 mg Selpercatinib: Participants received a single oral dose of 160 mg selpercatinib on Day 1 of Period 1.
- Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole: Participants received an oral dose of 200 mg itraconazole administered QD for 11 consecutive days (Days -4 to 7) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 of Period 2.
- Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin: Participants received an oral dose of 600 mg rifampin administered QD for 16 consecutive days (Days 1 to 16) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 of Period 2.
- Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin: Participants received an oral dose of 600 mg rifampin administered QD for 16 consecutive days (Days 1 to 16) with a single oral dose of 160 mg selpercatinib co-administered on Day 10 of Period 2.
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
nanogram *hour per milliliter (ng*h/mL) | 22380 (31.8) | 51570 (41.9) | 21070 (24.4) | 14080 (39.2) | 2784 (39.1)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Selpercatinib
Description: PK: AUC0-inf of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
ng*hr/mL | 22490 (31.4) | 52450 (41.6) | 21180 (23.9) | 16310 (33.4) | 2820 (38.9)

3. Primary Outcome: PK: Percentage of AUC0-inf Extrapolated (AUC%Extrap) of Selpercatinib
Description: PK: AUC%extrap of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf extrapolated
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
percentage of AUC0-inf extrapolated | 0.3377 (82.1) | 1.531 (48.1) | 0.3405 (98.9) | 12.33 (44.7) | 1.081 (67.9)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Description: PK: Maximum observed concentration (Cmax) of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
nanograms per milliliter (ng/mL) | 1442 (79.7) | 1880 (78.0) | 1364 (49.6) | 1624 (52.6) | 411.2 (40.3)

5. Primary Outcome: PK: Time to Reach Cmax (Tmax) of Selpercatinib
Description: PK: Tmax of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
hours (h) | 1.502 [1.00 to 24.01] | 1.502 [1.50 to 23.92] | 1.500 [1.00 to 8.03] | 2.003 [1.50 to 3.01] | 1.503 [1.00 to 2.50]

6. Primary Outcome: PK: Apparent First-order Terminal Elimination Rate Constant (Kel) of Selpercatinib
Description: PK: Kel of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
1/hour | 0.03428 (0.0047764) | 0.02493 (0.0026203) | 0.03567 (0.0080627) | 0.08861 (0.017055) | 0.06487 (0.021752)

7. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Selpercatinib
Description: PK: CL/F of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Mean (Standard Deviation); unit: Liters/hour
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
Liters/hour | 7.474 (2.8297) | 3.305 (1.5199) | 7.758 (1.9819) | 10.40 (4.5412) | 60.12 (20.457)

8. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Selpercatinib
Description: PK: t½ of Selpercatinib was reported.
  Outcome measure timeframe:
  Parts 1 and 2, Period 1: (Day 1) Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose.
  Part 1, Period 2; (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post dose. (contd.)
Time Frame: as for outcome 1
Population: All participants who received at least one dose of selpercatinib with evaluable PK data.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin | Part 2 Period 2: 160 mg Selpercatinib on Day 10 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12
h | 20.617 (3.1941) | 28.098 (3.0183) | 20.437 (5.1657) | 8.117 (1.7029) | 12.508 (6.2399)

9. Primary Outcome: Part 2 - PK: Area Under the Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24) of Selpercatinib Post Dose Day 1
Description: PK: AUC0-24 of Selpercatinib in Part 2 was reported.
Time Frame: Part 2, Periods 1 and 2: (Day 1) pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours post dose.
Population: All participants in Part 2 who received at least one dose of selpercatinib on Day 1 of either period with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib on Day 1 + 600 mg Rifampin
Number analyzed (Participants) | 12 | 12
ng*h/mL | 13240 (33.3) | 14090 (39.2)

ADVERSE EVENTS:
Time Frame: Baseline Up To 50 Days
Description: All participants who received at least one dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Per pre-specified analysis, adverse events were reported as per the treatment regimen received.
Groups:
- Part 2 Period 2: 160 mg Selpercatinib + 600 mg Rifampin: Participants received an oral dose of 600 mg rifampin administered QD for 16 consecutive days (Days 1 to 16) with a single oral dose of 160 mg selpercatinib co-administered on Day 1 and Day 10 of Period 2.
Arm/Group | Part 1 Period 1: 160 mg Selpercatinib | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole | Part 2 Period 1: 160 mg Selpercatinib | Part 2 Period 2: 160 mg Selpercatinib + 600 mg Rifampin
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 4/12 | 3/12 | 5/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1 Period 1: 160 mg Selpercatinib (N=12) | Part 1 Period 2: 160 mg Selpercatinib + 200 mg Itraconazole (N=12) | Part 2 Period 1: 160 mg Selpercatinib (N=12) | Part 2 Period 2: 160 mg Selpercatinib + 600 mg Rifampin (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear canal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (9)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0/6 (0) | 1/6 (1) | 0/5 (0) | 0/5 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT05338489/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/89/NCT05338489/SAP_001.pdf